CLINICAL TRIAL: NCT03148899
Title: Impact of Oxytocin on Obstructive Sleep Apnea Induced Changes in Sleep
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: George Washington University (Other)
Responsible Party: Principal Investigator, Vivek Jain, Principle Investigator, George Washington University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: GWU_IRB_041333
Record Dates: First submitted 2017-03-30; First posted 2017-05-11 (Actual); Results first posted 2023-01-31 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: Sleep Apnea, Obstructive
Keywords: Sleep Apnea; Oxytocin Nasal Spray
MeSH Terms: conditions — Sleep Apnea, Obstructive; Sleep Apnea Syndromes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: All members of the research team except the IP dispensing staff will be blinded for the duration of the research study. Once all the subjects have finished in the research study, and all data is data-locked, the outcomes assessor will then unblind the research data for the statistical analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Visit 1 Randomization (Experimental): At visit 1 (PSG 1) subjects will receive one of two interventions: either Oxytocin Intranasal Spray (40 IU) or Placebo Intranasal Spray. Subjects will be blinded as to which drug they are receiving.
  Interventions: Drug: Oxytocin Intranasal Spray; Drug: Placebo Intranasal Spray
- Visit 2: Crossover Randomization (Experimental): At visit 2 (PSG 2) subjects will receive the opposite intervention from the one they received at visit 1: either Oxytocin Intranasal Spray (40 IU) or Placebo Intranasal Spray. Subjects will be blinded as to which drug they are receiving.
  Interventions: Drug: Oxytocin Intranasal Spray; Drug: Placebo Intranasal Spray

INTERVENTIONS:
Drug: Oxytocin Intranasal Spray — In human volunteers intranasal administration of oxytocin significantly increases parasympathetic and decreases sympathetic cardiac control. In addition to the classic effects of oxytocin on uterine contraction and milk ejection, recent work indicates oxytocin is present in both males and females and has an important role in both behavior and cardiovascular homeostasis, particularly during anxiety and stress.
  Other Names: Synotocin
Drug: Placebo Intranasal Spray — The placebo has been compounded to be an inactive, blinded comparative to the oxytocin nasal spray.
  Other Names: Placebo

SUMMARY:
In human volunteers intranasal administration of oxytocin significantly increases parasympathetic and decreases sympathetic cardiac control. OSA is a very prevalent disease with high cardiovascular risk factors, yet this disease remains very poorly treated.

This proposal, based on the current literature and new basic science results detailed above on the role of oxytocin in cardiovascular control, will test if oxytocin administration improves adverse cardiovascular events during the recurrent nocturnal apneas in patients with OSA. This project will lay the groundwork and provide preliminary data to obtain NIH funding to test this important hypotheses more thoroughly and in larger clinical trials.

This study will explore if intranasal oxytocin has any positive cardiovascular benefits in patients with sleep apnea.

DETAILED DESCRIPTION:
Obstructive Sleep Apnea (OSA) is a major, yet poorly understood cardiovascular health risk that occurs in as many as 24% of males and 9% of females within the US population. OSA can participate in both the initiation and progression of several cardiovascular diseases including sudden death, hypertension, arrhythmias, myocardial ischemia and stroke.

Many of the adverse cardiovascular consequences of OSA are thought to be associated with a diminished cardiac vagal activity, as parasympathetic cardiac vagal activity is typically cardio-protective. Intranasal administration of oxytocin has been shown to significantly increase parasympathetic and decrease sympathetic cardiac control. In this research study, the effect oxytocin has on changes in heart rate or other Polysomnography (PSG) measures in a group of patients that have recently been diagnosed with OSA will be examined.

OSA is typically diagnosed through a polysomnography, a comprehensive recording of the biophysiological changes that occur during sleep. The PSG monitors many body functions including brain (EEG), eye movements (EOG), muscle activity or skeletal muscle activation (EMG) and heart rhythm (ECG) during sleep, respiratory airflow, respiratory effort, pulse oximetry etc.

In this research study, subjects who have recently been diagnosed with OSA will undergo two research study PSGs. Before the first study PSG, subjects will be randomized to receive either Oxytocin (40 IU) or placebo, in a blinded manner, prior to beginning the test. The PSG will then continue as usual, and subject data pertaining to the PSG will be gathered. Subjects will then return within 4 weeks for a second research PSG, where one hour before the test they will receive the opposite intervention that they did not received during the first research PSG study. Data measurements will be re-measured and compared between the two PSGs.

ELIGIBILITY:
Inclusion Criteria:

* Men or women 18 years old or older of any ethnic background
* Subjects that have recently undergone a standard "in the sleep-lab" diagnostic polysomnography (per standard of care medical guidelines), or the "at home" diagnostic test, and have been diagnosed with OSA

Exclusion Criteria:

* Pregnant or Breastfeeding women
* Women of Child Bearing Potential who are not willing to undergo methods to prevent pregnancy
* Subjects who are on medications that affect cardiac autonomic function (eg. Beta Blockers)
* Active smokers
* Subjects who are unable to read or answer questions in the English language

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2016-07-27 (Actual); Primary Completion 2020-06-07 (Actual); Study Completion 2020-06-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vivek Jain, MD, Principal Investigator — The George Washington University; David Mendelowitz, Principal Investigator — The George Washington University
Locations (1):
- The GW Medical Faculty Associates, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No
At this time there is no plan to share IPD

REFERENCES:
- [Derived] Jain V, Kimbro S, Kowalik G, Milojevic I, Maritza Dowling N, Hunley AL, Hauser K, Andrade DC, Del Rio R, Kay MW, Mendelowitz D. Intranasal oxytocin increases respiratory rate and reduces obstructive event duration and oxygen desaturation in obstructive sleep apnea patients: a randomized double blinded placebo controlled study. Sleep Med. 2020 Oct;74:242-247. doi: 10.1016/j.sleep.2020.05.034. Epub 2020 Jun 5. PMID 32862007

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 36 subjects with OSA were assessed for eligibility and willingness to participate in this double blinded cross over placebo-controlled trial. Four subjects declined to participate. The remaining 32 subjects were randomly assigned to receive either placebo (n=16) or oxytocin (n=16) in the first visit, then a washout period within 4 weeks, then the other intervention they did not receive in the second visit.
Groups:
- Experimental: Oxytocin, Then Placebo: At visit 1 (PSG 1) subjects first will receive Oxytocin Intranasal Spray (40 IU).
  Oxytocin Intranasal Spray: In human volunteers intranasal administration of oxytocin significantly increases parasympathetic and decreases sympathetic cardiac control. In addition to the classic effects of oxytocin on uterine contraction and milk ejection, recent work indicates oxytocin is present in both males and females and has an important role in both behavior and cardiovascular homeostasis, particularly during anxiety and stress.
  Then, at visit 2 (PSG 2), after a washout period of up to 4 weeks, they then received the Placebo Intranasal Spray: The placebo has been compounded to be an inactive, blinded comparative to the oxytocin nasal spray.
  Subjects were blinded as to which drug they received first.
- Experimental: Placebo, Then Oxytocin: At visit 1 (PSG 1) subjects first will receive the Placebo Intranasal Spray: The placebo has been compounded to be an inactive, blinded comparative to the oxytocin nasal spray.
  Then, at visit 2 (PSG 2), after a washout period of up to 4 weeks, they then received the receive Oxytocin Intranasal Spray (40 IU).
  Oxytocin Intranasal Spray: In human volunteers intranasal administration of oxytocin significantly increases parasympathetic and decreases sympathetic cardiac control. In addition to the classic effects of oxytocin on uterine contraction and milk ejection, recent work indicates oxytocin is present in both males and females and has an important role in both behavior and cardiovascular homeostasis, particularly during anxiety and stress.
  Subjects were blinded as to which drug they received first.
Period: Overall Study
Arm/Group | Experimental: Oxytocin, Then Placebo | Experimental: Placebo, Then Oxytocin
Started | 16 | 16
Completed | 16 | 16
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: There were 32 participants total, 16 in each arm.
Groups:
- Oxytocin, Then Placebo: At visit 1 (PSG 1) subjects will receive one of two interventions: either Oxytocin Intranasal Spray (40 IU) or Placebo Intranasal Spray. Subjects will be blinded as to which drug they are receiving.
  Oxytocin Intranasal Spray: In human volunteers intranasal administration of oxytocin significantly increases parasympathetic and decreases sympathetic cardiac control. In addition to the classic effects of oxytocin on uterine contraction and milk ejection, recent work indicates oxytocin is present in both males and females and has an important role in both behavior and cardiovascular homeostasis, particularly during anxiety and stress.
  Placebo Intranasal Spray: The placebo has been compounded to be an inactive, blinded comparative to the oxytocin nasal spray.
- Placebo, Then Oxytocin: At visit 2 (PSG 2) subjects will receive the opposite intervention from the one they received at visit 1: either Oxytocin Intranasal Spray (40 IU) or Placebo Intranasal Spray. Subjects will be blinded as to which drug they are receiving.
  Oxytocin Intranasal Spray: In human volunteers intranasal administration of oxytocin significantly increases parasympathetic and decreases sympathetic cardiac control. In addition to the classic effects of oxytocin on uterine contraction and milk ejection, recent work indicates oxytocin is present in both males and females and has an important role in both behavior and cardiovascular homeostasis, particularly during anxiety and stress.
  Placebo Intranasal Spray: The placebo has been compounded to be an inactive, blinded comparative to the oxytocin nasal spray.
- Total: Total of all reporting groups
Arm/Group | Oxytocin, Then Placebo | Placebo, Then Oxytocin | Total
Number analyzed (Participants) | 16 | 16 | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 16 | 16 | 32
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.8 (9.1) | 42.8 (9.1) | 42.8 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 7 | 14
  Male | 9 | 9 | 18
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 16 | 16 | 32
Body-mass Index [Mean (Standard Deviation); unit: kg/m^2] | 31.8 (8.7) | 31.8 (8.7) | 31.8 (8.7)

OUTCOME MEASURES:

1. Primary Outcome: Duration of Obstructive Events
Time Frame: Assessed on Visit 1- Day 1, Visit 2- Day 29
Measure: Mean (Standard Deviation); unit: seconds
Groups:
- Oxytocin: At visit 1 (PSG 1) subjects will receive one of two interventions: either Oxytocin Intranasal Spray (40 IU) or Placebo Intranasal Spray. Subjects will be blinded as to which drug they are receiving.
  Oxytocin Intranasal Spray: In human volunteers intranasal administration of oxytocin significantly increases parasympathetic and decreases sympathetic cardiac control. In addition to the classic effects of oxytocin on uterine contraction and milk ejection, recent work indicates oxytocin is present in both males and females and has an important role in both behavior and cardiovascular homeostasis, particularly during anxiety and stress.
  Placebo Intranasal Spray: The placebo has been compounded to be an inactive, blinded comparative to the oxytocin nasal spray.
- Placebo: At visit 2 (PSG 2) subjects will receive the opposite intervention from the one they received at visit 1: either Oxytocin Intranasal Spray (40 IU) or Placebo Intranasal Spray. Subjects will be blinded as to which drug they are receiving.
  Oxytocin Intranasal Spray: In human volunteers intranasal administration of oxytocin significantly increases parasympathetic and decreases sympathetic cardiac control. In addition to the classic effects of oxytocin on uterine contraction and milk ejection, recent work indicates oxytocin is present in both males and females and has an important role in both behavior and cardiovascular homeostasis, particularly during anxiety and stress.
  Placebo Intranasal Spray: The placebo has been compounded to be an inactive, blinded comparative to the oxytocin nasal spray.
Arm/Group | Oxytocin | Placebo
Number analyzed (Participants) | 19 | 19
seconds | 22.72 (4.59) | 24.66 (5.12)

2. Secondary Outcome: Respiratory Rate
Time Frame: Assessed on Visit 1- Day 1, Visit 2- Day 29
Measure: Mean (Standard Deviation); unit: breaths per minute
Arm/Group | Oxytocin | Placebo
Number analyzed (Participants) | 19 | 19
breaths per minute | 17.39 (3.50) | 16.69 (3.24)

3. Secondary Outcome: Incidence Proportion of Bradycardia
Description: Event-associated bradycardias were identified as a heart rate reduction of 5 bpm or more from the average heart rate during the 5 s preceding an event to the lowest heart rate either during an event or within 5 s immediately after an event.
  Incidence proportion, or risk, of bradycardia was calculated as follows: the number of events that resulted in bradycardia divided by the total number of events.
  This analysis was done using custom MATLAB (MathWorks) code to study heart rate and peripheral capillary oxyhemoglobin saturation (SPO2) before and after apnea and hypopnea events.
Time Frame: Assessed on Visit 1- Day 1, Visit 2- Day 29
Measure: Mean (Standard Deviation); unit: proportion of events
Arm/Group | Oxytocin | Placebo
Number analyzed (Participants) | 19 | 19
proportion of events | 0.08 (0.07) | 0.14 (0.07)

4. Secondary Outcome: O2 Minimum
Time Frame: Assessed on Visit 1- Day 1, Visit 2- Day 29
Measure: Mean (Standard Deviation); unit: % of Oxygen Saturation
Arm/Group | Oxytocin | Placebo
Number analyzed (Participants) | 19 | 19
% of Oxygen Saturation | 94.31 (1.80) | 92.44 (4.24)

ADVERSE EVENTS:
Time Frame: 6 weeks
Description: There were no adverse events.
Arm/Group | Oxytocin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/32
Other Adverse Events (participants affected / at risk) | 0/32 | 0/32

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan: Protocol w/ SAP (2017-12-14): https://cdn.clinicaltrials.gov/large-docs/99/NCT03148899/Prot_SAP_000.pdf